CLINICAL TRIAL: NCT05214989
Title: Development of a Tailored Intervention to Increase Veteran Enrollment in Cardiac Rehabilitation (CDA 19-391)
Brief Title: Tailored Interventions to Increase Cardiac Rehabilitation Enrollment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We obtained information that referral rates are very low across the VA system for cardiac rehabilitation services, rendering the proposed clinical trial obsolete. Further information is detailed in the RPPR for the associated Career Development Award
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDX 22-003
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Disease
Keywords: Cardiac Rehabilitation; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This is a single group proof of concept study of an intervention involving tailored counseling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tailored intervention (Experimental): Tailored intervention designed to address individual barriers to cardiac rehabilitation participation
  Interventions: Behavioral: Tailored intervention

INTERVENTIONS:
Behavioral: Tailored intervention — Tailored intervention designed to address individual barriers to cardiac rehabilitation participation

SUMMARY:
Cardiac rehabilitation, an outpatient program that includes supervised exercise and cardiovascular risk factor education, is one of the most important therapies for patients with cardiovascular disease. Unfortunately, very few Veterans with cardiovascular disease enroll in cardiac rehabilitation programs. This proposal will evaluate Veterans' individual barriers to attending cardiac rehabilitation with both surveys and interviews. Using this information, the investigators will develop a behavioral intervention to encourage Veterans to enroll in outpatient cardiac rehabilitation programs. This intervention will be individually tailored to Veterans with the information- motivation-behavioral skills model, a theory of behavior change. The investigators will test the tailored intervention with a proof-of-concept study in Veterans hospitalized with cardiovascular disease at the Veterans Affairs Tennessee Valley Healthcare System. This project is relevant to Veterans' health because increasing enrollment in cardiac rehabilitation will decrease mortality and increase quality of life in Veterans with cardiovascular disease.

DETAILED DESCRIPTION:
Background: This Veterans Affairs (VA) Health Services Research & Development Career Development Award resubmission is a five-year plan that will enable the candidate, a staff cardiologist and specialist in cardiac rehabilitation (CR) at the VA Tennessee Valley Healthcare System, to develop and implement interventions to increase CR enrollment in Veterans. CR is an outpatient program including prescriptive exercise and cardiac risk factor education that is an essential therapy for patients with cardiovascular disease. This proposal will develop a tailored intervention to increase Veteran enrollment in CR.

Significance/Impact: CR is widely underutilized, with less than 20% of eligible patients enrolling in CR programs nationally. CR utilization is particularly low among Veterans, with only 10% of eligible Veterans enrolling in CR programs. Though CR referral rates have risen substantially over the past decade, CR enrollment has remained static. It is imperative to study barriers to CR enrollment among Veterans that have already been referred to CR and develop interventions tailored to these individual barriers.

Innovation: The applicant will develop a tailored intervention for increasing CR enrollment using the Obesity- Related Behavioral Intervention Trials model, a conceptual model for intervention development, as well as the information-motivation-behavioral skills model, a theory of behavior change that allows individual tailoring. Linking these models will produce new knowledge regarding behavioral intervention methodology as well as an innovative clinical intervention that can be delivered by nurses and other clinical staff at VA facilities. The proposed intervention aligns with current VA initiatives by supporting CR enrollment wherever is most convenient for Veterans (including VA CR programs, non-VA CR programs, and home-based CR programs).

Specific Aims: Aims 1 and 2 comprise a sequential explanatory mixed methods study to evaluate barriers to CR enrollment among Veterans. The purpose of Aim 1 is to quantify barriers to CR in 100 Veterans hospitalized with ischemic heart disease using the previously validated Beliefs About Cardiac Rehabilitation Scale (BACRS). The purpose of Aim 2 is to reveal additional barriers to outpatient CR enrollment through qualitative interviews in 30 Veterans from Aim 1 who did not enroll in CR. Aim 3 focuses on the iterative development of a tailored intervention to increase outpatient CR enrollment in 3 groups of 5 hospitalized Veterans, characterizing the intervention's feasibility and acceptability. In Aim 4, the tailored intervention will undergo proof-of-concept testing in a non-randomized group of 25 Veterans hospitalized with ischemic heart disease. The applicant hypothesizes that these Veterans will have a clinically significant improvement in BACRS summary scores after the intervention, representing a decrease in perceived barriers to CR.

Methodology: Aim 1 will quantitate the burden of CR barriers among Veterans by evaluating distributions of BACRS summary scores and subscales. In Aim 2, the applicant will use intensity sampling to purposefully select Veterans with the lowest individual BACRS subscale scores (and highest perceived barriers to CR) from the Aim 1 cohort for semi-structured qualitative interviews. Aim 3 will use mixed data from Aims 1 and 2 and serial formative evaluations to inform the iterative development of a tailored intervention. In Aim 4, the BACRS will be administered before and after the intervention, characterizing the intervention's effect on perceived barriers to CR enrollment as measured by the BACRS summary score.

Implementation/Next Steps: The applicant will align the study activities with the QUERI Implementation Roadmap and convene a Stakeholder Engagement Panel to ensure that the tailored intervention is developed with maximum generalizability to other VA facilities. Findings from the proposed study will inform a wide range of initiatives related to CR enrollment among Veterans and will be used to conduct a randomized clinical trial of the tailored intervention within the context of an Investigator Initiated Research application.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients undergoing coronary artery bypass grafting or percutaneous coronary intervention.

Exclusion Criteria:

* Inability to communicate in English
* Blindness
* Hearing impairment
* Conditions that would interfere with the validity of the questionnaire (e.g., significant dementia, active psychosis or mania), being near the end of life (hospice or home hospice)
* Lack of cooperation
* Police custody
* Participation in a cardiac rehabilitation program within the previous year, or enrollment in a conflicting study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Qualitative interviews | 1-2 days after intervention
  Qualitative interviews will evaluate the effectiveness of the intervention in changing attitudes towards cardiac rehabilitation participation.

CONTACTS AND LOCATIONS:
Overall Officials: Justin M Bachmann, MD MPH, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (1):
- Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No